CLINICAL TRIAL: NCT04323644
Title: Outcomes of Surgery in COVID-19 Infection: International Cohort Study (CovidSurg)
Acronym: CovidSurg
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: CS-20200324
Record Dates: First submitted 2020-03-25; First posted 2020-03-26 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Coronavirus; Surgery
Keywords: COVID-19; Coronavirus; Surgery
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Patients with COVID-19 infection undergoing surgery
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Emergency or elective surgery

SUMMARY:
CovidSurg will capture real-world international data, to determine 30-day mortality in patients with COVID-19 infection who undergo surgery. This shared international experience will inform the management of this complex group of patients who undergo surgery throughout the COVID-19 pandemic, ultimately improving their clinical care.

DETAILED DESCRIPTION:
There is an urgent need to understand the outcomes of COVID-19 infected patients who undergo surgery. Capturing real-world data and sharing international experience will inform the management of this complex group of patients who undergo surgery throughout the COVID-19 pandemic, improving their clinical care.

The primary aim of the study is to determine 30-day mortality in patients with COVID-19 infection who undergo surgery. In doing so, this will inform future risk stratification, decision making, and patient consent.

CovidSurg is an investigator-led, non-commercial, non-interventional study is extremely low risk, or even zero risk. This study does not collect any patient identifiable information (including no dates) and data will not be analysed at hospital-level.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ANY type of surgery in an operating theatre, this includes obstetrics

AND

- The patient had COVID-19 infection either at the time of surgery or within 30 days of surgery, based on

(i) positive COVID-19 lab test or computed tomography (CT) chest scan

OR

(ii) clinical diagnosis (no COVID-19 lab test or CT chest performed)

Exclusion Criteria:

* If COVID-19 infection is diagnosed >30 days after discharge, the patient should not be included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with COVID-19 infection who undergo surgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  Death up to 30-days post surgery

SECONDARY OUTCOMES:
7-day mortality | 7 days post surgery
  Death up to 7-days post surgery
30-day reoperation | Up to 30-days post surgery
  Reoperation up to 30-days post surgery
Postoperative ICU admission | Up to 30 days post surgery
  Admission to ICU post surgery
Postoperative respiratory failure | Up to 30 days post surgery
  Respiratory failure post surgery
Postoperative acute respiratory distress syndrome (ARDS) | Up to 30 days post surgery
  Acute respiratory distress syndrome post surgery
Postoperative sepsis | Up to 30 days post surgery
  Sepsis post surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available to other researchers

REFERENCES:
- [Derived] COVIDSurg Collaborative. Outcomes after perioperative SARS-CoV-2 infection in patients with proximal femoral fractures: an international cohort study. BMJ Open. 2021 Nov 30;11(11):e050830. doi: 10.1136/bmjopen-2021-050830. PMID 34848515
- [Derived] Seeliger B, Philouze G, Cherkaoui Z, Felli E, Mutter D, Pessaux P. Acute abdomen in patients with SARS-CoV-2 infection or co-infection. Langenbecks Arch Surg. 2020 Sep;405(6):861-866. doi: 10.1007/s00423-020-01948-2. Epub 2020 Jul 27. PMID 32720012